CLINICAL TRIAL: NCT01901185
Title: A Single-arm, Multicenter Study to Evaluate the Ability of Subjects With Rheumatoid Arthritis or Psoriatic Arthritis to Effectively Use a Reusable Electromechanical Autoinjector to Self-inject Etanercept
Brief Title: Study to Evaluate the Ability of Subjects With Rheumatoid Arthritis or Psoriatic Arthritis to Effectively Use a Reusable Autoinjector to Self-inject Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110107
Record Dates: First submitted 2013-05-17; First posted 2013-07-17 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept / Autoinjector A (Experimental): Participants self-injected 50 mg etanercept subcutaneously using autoinjector A at the study center on Day 1 and then once a week from Weeks 1 to 5 (total of 6 injections).
  Interventions: Drug: Etanercept / Autoinjector A

INTERVENTIONS:
Drug: Etanercept / Autoinjector A — Autoinjector A, a hand-held, reusable electromechanical device, and a single-use, disposable cassette preassembled with an etanercept 50-mg liquid prefilled syringe (PFS).
  Other Names: Enbrel®

SUMMARY:
The purpose of this study is to assess the ability of people with rheumatoid arthritis (RA) or psoriatic arthritis (PsA) to use an experimental autoinjector to self inject etanercept (Enbrel®).

DETAILED DESCRIPTION:
Study participants need to have been self-administering etanercept for greater than or equal to 6 months prior to screening. You will be in this study for about 9 weeks. This includes a 4-week screening period and a 5-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of RA or PsA and indicated for treatment with etanercept per the current label, based on history.
* Subject is willing to self-inject per investigator judgement at screening.
* Subject has no known history of tuberculosis.

Exclusion Criteria:

* Latex allergy.
* Subject has any active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to first study dose of etanercept.
* Subject had prosthetic joint infection within 5 years of screening or native joint infection within 1 year of screening.
* Other criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2013-12-18 (Actual); Study Completion 2013-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (13):
  - Research Site, Huntsville, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Santa Maria, California
  - Research Site, Upland, California
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Paducah, Kentucky
  - Research Site, Lincoln, Nebraska
  - Research Site, Orchard Park, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with rheumatoid arthritis (RA) or psoriatic arthritis (psA) currently receiving treatment with etanercept were eligible to enrol in this study.
  First patient enrolled on 11 June 2013; last patient enrolled on 13 November 2013.
Period: Overall Study
Arm/Group | Etanercept / Autoinjector A
Started | 77
Received Etanercept With Autoinjector A | 75
Completed | 75
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept / Autoinjector A
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  White | 74
  Other | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 14
  Not Hispanic/Latino | 63
Disease state [Number; unit: participants]
  Rheumatoid arthritis | 66
  Psoriatic arthritis | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Successful Self-injections to Total Non-missed Injections
Description: The successful self-injection of etanercept using the Autoinjector A, as evaluated by the percentage of successful injections of the total nonmissed injections administered by participants in the non-health care setting during Weeks 1 to 5. Successful self-injection was assessed by Question 1 in the Participant Self-injection Questionnaire, which was completed by each participant after each self-injection. Successful injection is defined as the Autoinjector A signaling a complete injection and no liquid medication pooled on your skin.
Time Frame: Week 1, Week 2, Week 3, Week 4 and Week 5
Population: Primary analysis set defined as all nonmissed injections using Autoinjector A during Weeks 1 to 5 for all enrolled participants; in the event of multiple injection attempts, only the last attempt per week was counted.
Measure: Number (95% Confidence Interval); unit: percentage of successful injections
Units Other Than Participants: nonmissed injections
Arm/Group | Etanercept / Autoinjector A
Number analyzed (Participants) | 75
Number analyzed (nonmissed injections) | 367
percentage of successful injections | 97.8 [96.3 to 99.3]

2. Secondary Outcome: Percentage of Autoinjector A System Failures
Description: The autoinjector A and prefilled syringe (PFS)/cassettes used by the participants were examined at the end of the study by device engineers. System failure was defined as the failure of the Autoinjector A or PFS/cassette to meet the device design requirements during Weeks 1 to 5. The percentage of system failures is reported out of the total number of injection attempts during the study, including multiple attempts per week.
Time Frame: Week 1, Week 2, Week 3, Week 4 and Week 5
Population: Primary analysis set; multiple injection attempts per week are included.
Measure: Number (95% Confidence Interval); unit: percentage of system failures
Units Other Than Participants: total injection attempts
Arm/Group | Etanercept / Autoinjector A
Number analyzed (Participants) | 75
Number analyzed (total injection attempts) | 373
percentage of system failures | 2.4 [1.0 to 4.0]

3. Secondary Outcome: Percentage of Errors in Each Step of the Self-injection Process
Description: For all the nonmissed injections recorded on the Participant Self-injection Questionnaire, the percentage of the following steps in the self-injection process that were not successfully completed out of the total nonmissed injections during Weeks 1 to 5 are reported. If multiple attempts were recorded, all the recorded attempts were considered, regardless whether it was a successful attempt or not. • Error Icon lit up (Question 2) • Could not load cassette successfully (Question 3) • Could not remove purple cassette cap successfully (Question 4) • Could not press start button to begin self-injection successfully (Question 5).
Time Frame: Week 1, Week 2, Week 3, Week 4 and Week 5
Population: Primary analysis set; multiple injection attempts per week are included.
Measure: Number; unit: percentage of errors
Units Other Than Participants: total injection attempts
Arm/Group | Etanercept / Autoinjector A
Number analyzed (Participants) | 75
Number analyzed (total injection attempts) | 373
percentage of errors
  Error icon lit up | 4.3
  Could not load cassette successfully | 1.9
  Could not remove purple cassette cap successfully | 1.1
  Could not press start button to begin injection | 1.6

4. Other Pre Specified Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Adverse Device Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant that does not necessarily have a causal relationship with study treatment or the device under study. The definition includes worsening of a pre-existing medical condition. A serious adverse event is defined as an AE that meets at least 1 of the following serious criteria: • fatal • life threatening • requires or prolongs in-patient hospitalization • results in persistent or significant disability/incapacity • congenital anomaly/birth defect • other medically important serious event. An adverse device effect is any adverse event related to the use of a medical device. Adverse device effects include AEs resulting from insufficient or inadequate instructions for use, malfunction of the device, or from use errors (including errors resulting from normal use, reasonably forseeable misuse or from intentional misuse) of the device.
Time Frame: 9 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Etanercept / Autoinjector A
Number analyzed (Participants) | 75
participants
  All adverse events | 21
  Serious adverse events | 1
  Adverse events associated with device | 10

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Autoinjector A/Etanercept: Participants self-injected 50 mg etanercept subcutaneously using autoinjector A at the study center on Day 1 and then once a week at Weeks 1 - 5 (total of 6 injections).
Arm/Group | Autoinjector A/Etanercept
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 14/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autoinjector A/Etanercept (N=75)
Gastroenteritis viral (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autoinjector A/Etanercept (N=75)
Injection site pain (General disorders) | 12
Injection site reaction (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.